CLINICAL TRIAL: NCT00468091
Title: Regulation of Antro-pyloro-duodenal and Proximal Gastric Motility by GLP-1: Involvement of Cholinergic Pathways
Brief Title: Effects of Exendin(9-39) on Gastroduodenal Motility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Research Foundation (Other); Philipps University Marburg (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MATEX; DFG Ar149/1-2; DFG 527/5-2
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2007-04

CONDITIONS: Digestive Physiology; Gastrointestinal Motility; Gastrointestinal Hormones; Glucagon-like Peptide 1; Exendin (9-39)
Keywords: GLP-1; exendin(9-39); atropine; human; motility
MeSH Terms: interventions — exendin (9-39); Atropine

ARMS (4):
- saline-saline (Placebo Comparator): saline IV
  + saline IV
- saline-exendin(9-39)amide (Active Comparator): saline IV
  + exendin(9-39)amide IV
  Interventions: Drug: exendin(9-39)amide
- saline-atropine (Active Comparator): saline IV
  + atropine IV
  Interventions: Drug: atropine
- exendin(9-39)amide-atropine (Active Comparator): exendin(9-39)amide IV
  + atropine IV
  Interventions: Drug: exendin(9-39)amide; Drug: atropine

INTERVENTIONS:
Drug: exendin(9-39)amide
  Arms: exendin(9-39)amide-atropine; saline-exendin(9-39)amide
Drug: atropine
  Arms: exendin(9-39)amide-atropine; saline-atropine

SUMMARY:
The purpose of this study in humans is to define the effects of the endogenous hormone GLP-1 on gastroduodenal motility and on endocrine pancreatic secretion by using the specific GLP-1 receptor antagonist exendin(9-39). To elucidate possible cholinergic pathways, we combined exendin(9-39) with the muscarinergic antagonist atropine.

DETAILED DESCRIPTION:
Following a meal, gut-produced incretin hormones such as glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) are released into the circulation. GLP-1 and GIP, the two dominant incretin hormones, are part of a natural endogenous system involved in maintaining glucose homeostasis. In the presence of normal or elevated, but not low, glucose concentration, both GLP-1 and GIP increase insulin secretion from pancreatic islet beta-cells. GLP-1 also lowers glucagon secretion from pancreatic alpha-cells and delays nutrient delivery from the stomach by inhibiting gastric emptying. These combined effects improve glucose tolerance providing the rationale for a therapeutic potential of GLP-1 analogues in the treatment of diabetes mellitus.

A dominant gastrointestinal action of synthetic GLP-1 is the inhibition of gastroduodenal and stimulation of pyloric motility, resulting in a delay of gastric emptying and in decreased glycemic excursions. Postprandial glucose fluctuations have been demonstrated to be an important determinant of glycemic control as assessed by A1C. Moreover, emerging evidence shows a strong link between transient postprandial hyperglycemia and microvascular and macrovascular complications in diabetes mellitus. Deceleration of gastric emptying is now considered as mechanism to lower postprandial glycemia in patients with diabetes mellitus. It is part of the pharmacodynamic profile of new antidiabetic incretinomimetica. In contrast, inhibition of the enzyme dipeptidylpeptidase 4 (DPP-4) which is responsible for the rapid degradation of GLP-1 failed to show an effect on gastric emptying in human although plasma GLP-1 was increased by twofold. Most of our understanding of the effects of GLP-1 is based upon studies employing synthetic GLP-1 whereas only little is known about endogenously released GLP-1.

Using the specific GLP-1 receptor antagonist exendin(9-39) we were able to show that endogenous GLP-1 acts as an incretin hormone in human. Moreover, the inhibition of antroduodenal and the stimulation of pyloric motility during a duodenal glucose load were reversed by the GLP-1 receptor antagonist. In order to more completely evaluate the effects of GLP-1 as an enterogastrone, the present study examines the effects of exendin(9-39) on antropyloroduodenal and proximal gastric motility during a physiological meal. As cholinergic pathways are thought to be involved in inhibitory actions of GLP-1 we combine the GLP-1 receptor antagonist with the muscarinergic antagonist atropine. To ensure a comparable stimulation of GLP-1 under all experimental conditions we decide to perfuse the meal directly into the duodenum.

Comparisons: In ten healthy volunteers, an interdigestive period is followed by 70 min with duodenal perfusion of a mixed liquid meal (250 kcal). On four days and in random order, exendin(9-39) (300 pmol•kg-1•min-1), atropine (5 µg•kg-1•h-1), exendin(9-39) + atropine or saline are intravenously infused. Antro-pyloro-duodenal perfusion manometry and fundic motility (electronic barostat) are assessed in parallel. Isobaric distensions of the proximal stomach were performed determining compliance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (postmenopausal, surgically sterile or using double-barrier method of contraception) healthy volunteers
* Age 18-65 years
* Body mass index (BMI) < 30 kg/m2
* Must have a fasting blood glucose below 100 mg/dl at screening and on all study days
* Able to provide written informed consent prior to study participation
* Able to communicate well with the investigator and comply with the requirements of the study

Exclusion Criteria:

* Diabetes mellitus
* Treatment with systemic steroids and thyroid hormone
* Patients with any history of gastrointestinal surgery, e.g. partial bowel resections, partial gastric resections, etc.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Past medical history of clinically significant electrocardiogram (ECG) abnormalities or a family history of a prolonged QT-interval syndrome.
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study. The investigator should be guided by evidence of any of the following:
* history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding
* history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
* history or clinical evidence of pancreatic injury or pancreatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1999-02; Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Effect of exendin(9-39) on gastroduodenal motility Effect of exendin(9-39) on gastroduodenal motility with simultaneous atropine | within the 200 min study period

SECONDARY OUTCOMES:
Effect of exendin(9-39) on blood glucose levels and plasma immunoreactivities of insulin, glucagon, and pancreatic polypeptide | within the 200 min study period

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schirra, MD, Principal Investigator — Clinical Research Unit, Dept. of Internal Medicine II, University of Munich
Locations (1):
- Clinical Research unit, Dept. of Internal Medicine II - Großhadern, University of Munich, Munich, Germany

REFERENCES:
- [Background] Schirra J, Sturm K, Leicht P, Arnold R, Goke B, Katschinski M. Exendin(9-39)amide is an antagonist of glucagon-like peptide-1(7-36)amide in humans. J Clin Invest. 1998 Apr 1;101(7):1421-30. doi: 10.1172/JCI1349. PMID 9525985
- [Background] Schirra J, Houck P, Wank U, Arnold R, Goke B, Katschinski M. Effects of glucagon-like peptide-1(7-36)amide on antro-pyloro-duodenal motility in the interdigestive state and with duodenal lipid perfusion in humans. Gut. 2000 May;46(5):622-31. doi: 10.1136/gut.46.5.622. PMID 10764704
- [Background] Schirra J, Wank U, Arnold R, Goke B, Katschinski M. Effects of glucagon-like peptide-1(7-36)amide on motility and sensation of the proximal stomach in humans. Gut. 2002 Mar;50(3):341-8. doi: 10.1136/gut.50.3.341. PMID 11839712
- [Background] Schirra J, Nicolaus M, Roggel R, Katschinski M, Storr M, Woerle HJ, Goke B. Endogenous glucagon-like peptide 1 controls endocrine pancreatic secretion and antro-pyloro-duodenal motility in humans. Gut. 2006 Feb;55(2):243-51. doi: 10.1136/gut.2004.059741. Epub 2005 Jun 28. PMID 15985560